CLINICAL TRIAL: NCT07202455
Title: Effect of Early Neuromodulation Coupled With Rehabilitation on the Prevention of Post-stroke Pain
Acronym: ENADA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RBHP 2025 MOISSET 2; 2025-A00988-41 (Other: 2025-A00988-41)
Record Dates: First submitted 2025-09-16; First posted 2025-10-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Neuropathic Pain; Central Post Stroke Pain
Keywords: neuropathic pain; prevention; stroke; central post stroke pain; neuromodulation; tDCS
MeSH Terms: conditions — Stroke; Neuralgia

STUDY DESIGN:
Intervention Model Description: Fleming plan (40 patients in the active group, 20 in the control group)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): Patients will receive 10 sessions of active tDCS stimulation (2mA, 20 minutes, 0.1mA/s ramp-up and ramp-down), in addition to conventional rehabilitation.
  Interventions: Device: Active tDCS
- Control group (Sham Comparator): Patients will receive 10 sessions of sham tDCS stimulation (2mA, 20 minutes, 0.1mA/s ramp-up, stimulation stopped after the current ramp), in addition to conventional rehabilitation.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Patients will receive 10 sessions of tDCS stimulation (2mA, 20 minutes with a current on/off ramp of 0.1 mA/s) delivered with a Sooma DUO stimulator. Sooma DUO is a transcranial direct current stimulation (tDCS) device. The device generates a current that modulates brain activity. This current is delivered via electrodes attached to the patient's head.
  Arms: Active group
Device: Sham tDCS — Patients will receive 10 sessions of sham tDCS stimulation (2mA, 20 minutes, 0.1mA/s ramp-up, stimulation stopped after the current ramp), delivered with a Sooma DUO stimulator. Sooma DUO is a transcranial direct current stimulation (tDCS) device. The device generates a current that modulates brain activity. This current is delivered via electrodes attached to the patient's head.
  Arms: Control group

SUMMARY:
This is a prospective clinical study to evaluate the efficacy of tDCS stimulation, coupled with conventional rehabilitation, on the development of post-stroke neuropathic pain.

The study involves a double-blind, randomized, sham-controlled experimental protocol involving 2 parallel groups with patients allocated according to a Fleming design (40 patients in the active group, 20 patients in the control group).

The study is aimed at sub-acute post-stroke patients. After recruitment, they will receive 10 sessions of tDCS stimulation (2mA, 20 minutes with a current on/off ramp of 0.1 mA/s). For the control group, stimulation will stop after the current ramp.

DETAILED DESCRIPTION:
Selection: during hospitalization in the neurology department of Clermont-Ferrand University Hospital, the principal investigator will propose that eligible patients take part in the ENADA study. If the patient agrees, an inclusion visit (E1) will be scheduled by the inclusion center. All these patients will have had an MRI recording as part of routine post-stroke practice.

Inclusion (E1 visit): A new background check and inclusion/non-inclusion criteria will be carried out. Once the patient has signed the study consent form, he or she will complete the self-questionnaires (VAS pain intensity, VAS pain affectivity, DN4, NPSI, BPI, HAD, diagram showing hypoesthetic areas, EQ-5D). The evaluation will also include FMA-UE test, the modified Ashworth scale and sensory thresholds.

Randomization: Patients will be randomized to the active or placebo group.

Protocol: 10 stimulation sessions, spread over a maximum of 21 consecutive working days.

Active and sham tDCS sessions are identical, double-blind. Stimulation by tDCS takes place during a physiotherapy, occupational therapy or speech therapy session. After installation, stimulation lasts 20 minutes. Stimulation is delivered at an intensity of 2 mA, with a ramp for the onset and disappearance of the current. Sham stimulation stops after the onset ramp, ensuring blindness for the patient, who may feel a slight tingling sensation during this phase. Patients will complete a pain intensity VAS and an affective pain VAS before and after each tDCS stimulation.

Post-protocol visit (visit E2): this visit is scheduled 7 days after the 10th and last stimulation session. It is carried out by the principal investigator at Clermont-Ferrand University Hospital.

An MRI recording is scheduled for this visit. Patients will fill in follow-up self-questionnaires (pain intensity VAS, affective pain VAS, DN4, NPSI, BPI, HAD, diagram showing hypoesthetic areas, EQ-5D), as well as their overall impression of change (PGIC score) and their impression of change on motor and sensory aspects. The evaluation will also include FMA-UE test and the modified Ashworth scale. The quality of blinding will be assessed at visit E2 by asking the patient's impression of the treatment he or she has received and of the presumed allocation (Bang blinding index).

End-of-study visit (E3 visit): this visit is scheduled at 6 months post-stroke. It is conducted by the principal investigator at the Clermont-Ferrand University Hospital.

The same assessments are carried out as at the previous visit, as well as the evaluation of sensory thresholds. In addition, the presence of neuropathic pain (yes/no), the primary endpoint, was assessed after clinical and instrumental evaluation. The presence of non-neuropathic pain (yes/no) is also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Ischemic or hemorrhagic stroke confirmed by MRI or scanner
* Lesion(s) in somato-sensory areas (i.e. mainly in: the pons, thalamus, internal capsule, basal ganglia and operculo-insular regions)
* Sensory and/or motor deficit requiring rehabilitation
* Subacute stage (7 to 45 days post-stroke)
* No neurological deficit or chronic neuropathic pain prior to stroke
* No neuropathic pain at inclusion
* Patient can be followed throughout the study.
* Information letter read and understood
* Able to give informed consent to participate in research
* Affiliation with a social security scheme

Exclusion Criteria:

* Contraindication to tDCS (epilepsy/history of epilepsy, intracranial ferromagnetic material or implanted stimulator, acute eczema or irritated skin over the stimulation area)
* Contraindication to MRI (use of a pacemaker or insulin pump, wearing of a metal prosthesis, intracerebral clip or piercing, claustrophobia)
* Cognitive or language difficulties preventing comprehension of instructions and/or correct clinical assessment
* Patients participating in another research protocol involving a drug in the 30 days prior to inclusion
* Drug or psychoactive substance abuse
* Pregnant or breast-feeding women
* Patients under guardianship or curatorship, deprived of liberty, safeguard of justice
* Major depression
* Patients with Parkinson's disease
* The presence of pre-existing lesions >1.5 cm (maximum diameter) in a cerebral area belonging to the anatomically defined sensorimotor system
* Alcohol abuse
* Severe psychiatric disorders (e.g., schizophrenia)
* Any tumor disease with a life expectancy of <1 year
* Increased intracranial pressure
* Patients with a medical device containing electronics or conductive materials
* Patients on continuous oxygen (system not adapted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Development of neuropathic pain | At 6 months post-stroke
  The primary endpoint is the development (yes/no) of probable or definite neuropathic pain according to IASP criteria, after clinical and instrumental assessment, at 6 months post-stroke.
  The presence of definite neuropathic pain will be recorded in the presence of negative sensory signs, i.e. partial or complete loss of one or more sensory modalities (e.g. light touch, cold temperature, etc.) concordant with the lesion of the somatosensory nervous system (in this case stroke, the presence of which will have been confirmed by MRI).

SECONDARY OUTCOMES:
Development of non-neuropathic pain | At 6 months post-stroke
  shoulder or other joint pain, spasticity-related pain, etc.
Pain intensity | Before the protocol, within 15 minutes before and after each tDCS session, after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Numeric Rating Scale (NRS) ranging from 0 (no pain) to 100 (worst pain imaginable)
Affective pain experience | Before the protocol, within 15 minutes before and after each tDCS session, after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Numeric Rating Scale (NRS) ranging from 0 (no affective impact of pain) to 100 (worst affective impact of pain)
Presence of neuropathic pain | Before and after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Douleur Neuropathique en 4 questions (DN4)
Evaluation of neuropathic pain | Before and after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Questionnaire d'évaluation des douleurs neuropathiques (NPSI)
Pain assessment | Before and after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Questionnaire concis sur les douleurs (BPI)
Motor function | Before and after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Fugl-Meyer Assessment - Upper extremity (FMA-UE) test, ranging from 0 (worst motor function) to 66 (correct motor function)
Spasticity | Before and after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Modified Ashworth Scale (MAS), ranging from 0 (no increase in muscle tone) to 4 (affectied part rigid in flexion or extension)
Anxiety and depression | Before and after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Hospital Anxiety and Depression (HAD) scale, ranging from 0 (no symptoms) to 21 (most severe symptoms)
Quality of life EQ-5D | Before and after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  EQ-5D scale, each item coded from 1 (no problem) to 3 (extreme problem)
Patient's impression of change | After the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Patient's global impression of change, impression of change in motor and sensory aspects, ranging from 1 (very significantly improved) to 7 (very significantly worsened)
Perceptual and pain hot and cold thresholds | Before the protocol and at six months post-stroke
  Thermal thresholds evaluated with a Thermotest, in the area with the most pronounced sensory symptoms and the contralateral similar area
Bang Blinding Index | After the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  Patient's impression of being in the active or control group, each patient report his/her impression (active group/control group/don't know) and proportions are compared between the active and control group
Brain activity | Before and after the protocol (within 7 days after the 10th and final tDCS session) and at six months post-stroke
  resting-state fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Moisset, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU Clemront-Ferrand, Clermont-Ferrand
  - CH Etienne Clémentel, Enval

IPD SHARING:
Plan to Share IPD: No